CLINICAL TRIAL: NCT01770314
Title: Medication Safety Pilot Study
Brief Title: Study to Test the Efficacy of Online Education to Increase Safe Use of Opioid Medication.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Inflexxion, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MedSafetyStudy; Endo Pharmaceuticals (Other: Endo Pharmaceuticals)
Record Dates: First submitted 2013-01-11; First posted 2013-01-17 (Estimated); Results first posted 2014-05-19 (Estimated); Last update posted 2014-05-19 (Estimated); Status verified 2014-04

CONDITIONS: Medication Adherence
Keywords: Opioid Pain Medication; Medication Safety; Correct storage; Correct disposal; Correct Use
MeSH Terms: conditions — Medication Adherence

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental (Experimental): Participants will be given instructions via email to review eleven online lessons about opioid medication safety. Instructions will suggest that participants view one lesson per day for eleven consecutive days. Each educational lesson focuses on one or two aspects of medication safety, including how to safely store medication, and the importance of taking medication exactly as prescribed.
  Interventions: Behavioral: Experimental
- Control (No Intervention): The control group is a waitlist control. Participants will be given access to painACTION after the intervention period and follow up assessments are completed.

INTERVENTIONS:
Behavioral: Experimental — Participants will be given instructions via email to review eleven online lessons about opioid medication safety. Instructions will suggest that participants view one lesson per day for eleven consecutive days. Each educational lesson focuses on one or two aspects of medication safety, including how to safely store medication, and the importance of taking medication exactly as prescribed.
  Other Names: painACTION website
  Arms: Experimental

SUMMARY:
The purpose of this project is to test whether an online pain medication intervention is a feasible and effective way to increase opioid pain medication safety.

DETAILED DESCRIPTION:
The goal of the study is to test the efficacy of the pain medication safety intervention for increasing safe management of prescription medication opioids. The study will use a randomized, controlled design that compares the intervention (painACTION medication safety lessons) to a waitlist control condition.

The hypotheses related to efficacy are that, as compared to the control group, people in the experimental group will demonstrate:

1. Increased self-efficacy for how to safely manage medications (primary outcome)
2. Increased behaviors associated with safely managing medication (secondary outcome)

Participants:

Investigators will recruit the first 148 respondents who meet the inclusion criteria and consent to be in the study.

Experimental Group. Participants will be given instructions via email to review eleven online lessons about opioid medication safety. Instructions will suggest that participants view one lesson per day for eleven consecutive days. Each educational lesson focuses on one or two aspects of medication safety, including how to safely store medication, and the importance of taking medication exactly as prescribed.

Control Group. The control group is a waitlist control. Participants will be given access to painACTION after the intervention period and follow up assessments are completed.

Randomization: Participants will be randomized by gender and age.

Procedure: Participants will be recruited with the help of the participating clinic. Staff members will let people know about the study by giving out informational fliers. The flier will direct people who are interested in participating in the study to an online screener. Those who screen in will automatically be lead to a consent form. Participants randomized to use painACTION will be sent the link to the online program and provided with a code that will serve as a Personal Identification Number (PIN) to access the program and return for subsequent sessions. The codes will also allow research staff to track program activity. The numbers are generated as participants agree to participate in the study and will begin with 0001 and continue to 0140 as the investigators add participants. The Research Coordinator will only provide assistance with the technical aspects of navigating the program. All assessments will be administered online. The battery will take no more than thirty minutes to complete. Several studies have determined that online assessments have many advantages over other modes of data collection (Webb et al., 1999; Yun, 2000). Online administration allows: (1) automation of the data collection process; (2) standardization of administration; (3) the use of personalized e-mail invitations at the precise assessment time points; (4) opportunities for participants to complete questionnaires on their own time and in the setting most comfortable to them; and (5) greater protection of confidentiality and conservation of resources because no written record exists. In addition, a number of studies have demonstrated that participants prefer computer-assisted self-interviews to traditional methods of data collection, and are more honest with computers (Johnston & Walton, 1995, Paperny et al., 2000). The increase in precision translates to greater power to detect real effect differences and higher confidence in the validity of the data. Information will not be saved if the browser is closed and the questionnaire has not been completed and submitted.

Assessments: Data will be collected from participants at baseline, immediately after the intervention, and one month post intervention.

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to provide consent
* Have the ability to read and write English
* Diagnosis of non-cancer chronic pain
* Prescribed opioids and taking consistently for 3 months.
* Over 18 years old

Exclusion Criteria:

* Previously visited painACTION

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2012-09; Primary Completion 2013-04 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Donovan, Ph. D., Principal Investigator — Inflexxion, Inc.
Locations (1):
- Inflexxion Inc, Newton, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited via an online advertisement as well as through posters
Groups:
- Control: The control group was a waitlist control. Participants were given access to the experimental intervention program after the intervention period and follow up assessments were completed.
- Experimental: Participants were given instructions via email to review eleven online lessons about opioid medication safety. Instructions suggested that participants view one lesson per day for eleven consecutive days. Each educational lesson focused on one or two aspects of medication safety, including how to safely store medication, and the importance of taking medication exactly as prescribed.
Period: Overall Study
Arm/Group | Control | Experimental
Started | 86 | 90
Contributed Data to Baseline | 68 | 72
Contributed Data to Post-test | 65 | 67
Contributed Data to One-month Follow-up | 61 | 66
Completed | 86 | 90
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental | Control | Total
Number analyzed (Participants) | 90 | 86 | 176
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 83 | 85 | 168
  >=65 years | 7 | 1 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 47 (11.8) | 45 (10.5) | 46 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 55 | 112
  Male | 33 | 31 | 64
Region of Enrollment [Number; unit: participants]
  United States | 90 | 86 | 176

OUTCOME MEASURES:

1. Primary Outcome: Self-efficacy - 8 Item Measure Taps Into Key Concepts Associated With Confidence for Managing Opioid Medications
Description: Responses are measured on a 4-point Likert scale (1= "Not at all confident" and 4= "Extremely confident"). The total Score range:8=least confident, 32=most confident.
  How confident do you feel in your ability to do each of the following activities, today?
  1. I can recognize side effects that are related to my opioid medicine.
  2. I can avoid giving my opioid medicine to someone else. Etc.. 1 - Not at all confident 2 - Somewhat confident 3 - Very confident 4 - Extremely confident Items have been generated from literature. Content validity: assessed by asking two experts if items are important and relevant.
  Internal consistency of the items in the pilot measure will be assessed (Cronbach's alpha).
  Test-retest reliability will be explored by asking 50 participants in the control group to retake the pilot measure within 3-5 days of having taken the measure as part of the pretest.
Time Frame: Baseline - Day 1, Posttest - Day 16 (intervention took 15 days), One month Followup - at 1 month post-intervention
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Experimental | Control
Number analyzed (Participants) | 90 | 86
units on a scale
  Baseline Least Square Means (n=72, 68) | 28.1081 (0.5412) | 27.0563 (0.5525)
  Post-test Least Square Means (n=67,65) | 29.7143 (0.4222) | 28.3224 (0.4254)
  One-month follow-up Least Square Means (n=66,61) | 30.2064 (0.4246) | 28.5664 (0.4352)

2. Secondary Outcome: Satisfaction With the Program
Description: We tested and analyzed participants' satisfaction with the program by asking the question: "Overall, how satisfied were you with the lessons." They answered on a 4 point Likert scale: 1=Not at all satisfied, 2=Somewhat Satisfied, 3=Satisfied, 4 = Very satisfied. Higher values indicate higher satisfaction.
Time Frame: One-month followup assessment
Population: We only analyzed satisfaction data for experimental participants who had indicated that they disposed of their unused opioid medications (n=17)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Experimental | Control
Number analyzed (Participants) | 17 | 0
units on a scale | 3.6470588 (0.6063391) |

ADVERSE EVENTS:
Arm/Group | Experimental | Control
Serious Adverse Events (participants affected / at risk) | 0/90 | 0/86
Other Adverse Events (participants affected / at risk) | 0/90 | 0/86

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes